CLINICAL TRIAL: NCT06229067
Title: Efficacy and Safety of PD-L1 Monoclonal Antibody Combined With Metronomic Chemotherapy of Vinorelbine, Cyclophosphamide and Capecitabine (VEX) Regime in Advanced Triple-negative Breast Cancer: a Multicenter, Randomized, Phase II Study
Brief Title: Efficacy and Safety of PD-L1 Monoclonal Antibody Combined With Metronomic VEX in Advanced Triple-negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Dr, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4279
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: PD-L1 inhibitor; immunotherapy; metronomic chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Vinorelbine; Cyclophosphamide; Tablets; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adebrelimab + VEX (Experimental): Adebrelimab at a dose of 1200 mg via intravenous infusion every three weeks, in combination with metronomic oral vinorelbine 20 mg every other day + cyclophosphamide 50 mg daily + capecitabine 500 mg three times daily
  Interventions: Drug: Adebrelimab; Drug: Vinorelbine; Drug: Cyclophosphamide (tablet); Drug: Capecitabine
- VEX (Active Comparator): Metronomic oral vinorelbine 20 mg every other day + cyclophosphamide 50 mg daily + capecitabine 500 mg three times daily
  Interventions: Drug: Vinorelbine; Drug: Cyclophosphamide (tablet); Drug: Capecitabine

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab at a dose of 1200 mg via intravenous infusion every three weeks. Adebrelimab will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
  Arms: adebrelimab + VEX
Drug: Vinorelbine — Metronomic oral vinorelbine 20 mg every other day. Vinorelbine will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
Drug: Cyclophosphamide (tablet) — Metronomic oral cyclophosphamide 50 mg daily. Cyclophosphamide will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.
Drug: Capecitabine — Metronomic oral capecitabine 500 mg three times daily. Capecitabine will continue to be administered as long as patient experiences clinical benefit in the opinion of the investigator or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data and clinical status or withdrawal of consent.

SUMMARY:
In recent years, immune therapy has significantly altered the treatment landscape for various malignant tumors, including breast cancer. Apart from its direct cytotoxic effects on tumor cells, metronomic chemotherapy has the potential to modulate the immune microenvironment, thereby demonstrating substantial synergistic potential with immune therapy. In a previous prospective adaptive randomized phase II clinical trial, we identified a promising regimen involving PD-1 monoclonal antibody in combination with vinorelbine + cyclophosphamide + capecitabine (VEX) metronomic chemotherapy. Building on this foundation, we plan to conduct a multicenter, randomized, controlled phase II study to evaluate the efficacy and safety of the PD-L1 monoclonal antibody in combination with VEX metronomic chemotherapy for patients with advanced triple-negative breast cancer, aiming to provide crucial evidence to guide medication for patients in advanced stages. The control group will receive metronomic oral vinorelbine 20 mg every other day + cyclophosphamide 50 mg daily + capecitabine 500 mg three times daily. The experimental group will receive additional PD-L1 inhibitor adebrelimab at a dose of 1200 mg via intravenous infusion every three weeks. Each cycle consists of three weeks, with imaging examinations conducted every six weeks (two cycles) to assess treatment efficacy. Subjects will continue medication until imaging indicates disease progression, toxicity becomes intolerable, withdrawal of informed consent, or the investigator deems it necessary to terminate medication. Evaluation will include efficacy indicators such as median progression-free survival, safety indicators like drug-related adverse reactions, patient survival quality, along with an exploratory analysis of biomarkers potentially associated with efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged ≥18 years who have signed informed consent and have an expected survival of ≥3 months.
2. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2 within 21 days prior to the first dose of medication.
3. Participants with clear clinical records of metastatic triple-negative breast cancer, as specified in the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines.
4. Participants with metastatic breast cancer who have received no more than first-line chemotherapy.
5. Participants with at least one measurable lesion, as defined by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
6. Participants with a history of receiving anthracycline and/or taxane-based treatments, including:

   1. Use of anthracyclines and/or taxanes during adjuvant or neoadjuvant therapy before breast cancer recurrence.
   2. Ineffectiveness observed during or after chemotherapy based on anthracyclines and/or taxanes.
   3. Participants deemed unsuitable for first-line treatment with anthracycline and/or taxane-based chemotherapy according to the investigator's judgment.
7. Completion of radiotherapy before the first dose of study medication, with a minimum interval of 4 weeks since the end of radiotherapy.
8. For participants with a history of surgery, a minimum interval of 30 days between surgery and the first dose of medication, with complete recovery from the surgical procedure.
9. Normal bone marrow function, evidenced by:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm².
   2. Platelets ≥ 100,000/mm².
   3. Hemoglobin (Hb) ≥ 10 g/dL.
10. Normal liver function, evidenced by:

    1. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN).
    2. Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 ULN (≤ 5.0 times ULN in the presence of liver metastasis).
    3. Alkaline phosphatase < 5 x ULN.
11. Normal renal function, evidenced by a creatinine clearance rate > 40 mL/min (Cockcroft-Gault formula).
12. Negative pregnancy test results within 7 days prior to the first dose of medication for women of childbearing potential, who also agree to employ necessary contraceptive measures.
13. Ability to understand and voluntarily sign the informed consent form before any study-related assessments/procedures.
14. Willingness and ability to comply with the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Current or past history of malignancies other than breast cancer, excluding: cured non-melanoma skin cancer, cured cervical carcinoma in situ, or cured other primary solid tumors with no evidence of disease activity and no curative treatment within the last 3 years.
2. Solely having pleural effusion, ascites, bone metastases, or other unmeasurable lesions.
3. Malabsorption syndrome or diseases significantly affecting gastrointestinal function, prior gastrectomy, or resection of the proximal small intestine that may affect the absorption of oral chemotherapeutic agents.
4. Swallowing difficulties or inability to swallow tablets.
5. Symptomatic brain or leptomeningeal metastasis; suspected signs or symptoms of central nervous system (CNS) involvement should be excluded by CT or MRI scans.
6. Other severe diseases or medical conditions discovered by the investigator during screening, including:

   1. Clinically significant heart diseases.
   2. Unstable diabetes.
   3. Uncontrolled hypercalcemia.
   4. Clinically significant active infections within the last 2 weeks.
7. History of organ transplantation.
8. Peripheral neuropathy of grade ≥2 according to NCI version 5.0.
9. Concurrent use of any other antitumor therapy for metastatic breast cancer.
10. Requirement for concurrent anticoagulant therapy.
11. Status of pregnancy, lactation, or unwillingness to use effective contraception for at least one month during the entire study period and for at least one month after the last dose of the study drug.
12. Known history of neurologic or psychiatric disorders or diseases that could compromise treatment compliance.
13. Less than a 3-week interval between the end of previous chemotherapy and the first dose of study medication.
14. Progressive disease during or after oral investigational drug treatment.
15. Use of any investigational drug within 30 days before starting study treatment. Less than 30 days since the use of any other investigational drug or device.
16. Known allergy to any component of the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-01-19 (Estimated); Primary Completion 2025-01-19 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 24 months
  Measured from the date of study drugs start to the date of the first objective disease progression or death.

SECONDARY OUTCOMES:
Overall Survival | 24 months
  Defined as the duration of time from start of treatment to time of death.
Disease Control Rate | 6 weeks of treatment
  Defined as the percentage of complete response (CR), partial response (PR) or stable Disease (SD). Response will be evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) V1.1.
Objective Response Rate | 6 weeks of treatment
  The objective response rate (ORR) will be defined as the proportion of patients described on the efficacy-evaluable population) who achieve complete response (CR) or partial response (PR) as best overall response at 6 weeks of treatment. ORR is based on tumor assessments.
Duration of Response | 24 months
  The length of time that a patient's disease remains in complete or partial remission after a response to treatment.
Adverse Events | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0